CLINICAL TRIAL: NCT06149728
Title: Pain Assessment and Transcranial Magnetic Stimulation Tolerability in Patients With a Functional Neurological Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Explorations Fonctionnelles Avicenne (Network)
Responsible Party: Principal Investigator, Ng Wing Tin, MD PhD, Explorations Fonctionnelles Avicenne
Other Study IDs: CLEA-2023-n°338
Record Dates: First submitted 2023-11-15; First posted 2023-11-29 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Functional Neurological Disorder
Keywords: Functional Neurological Disorder; Pain; TMS
MeSH Terms: conditions — Conversion Disorder; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Functional neurological disorders (FND) are motor, sensory or cognitive symptoms without an identified lesion. This is a very common reason for consultation in neurology. Transcranial magnetic stimulation (TMS) may be performed in these patients both for diagnostic purposes (in the context of motor evoked potentials) and for therapeutic purposes. The main objective of the study is to evaluate tolerability of TMS in patients with FND, in particular the pain caused by stimulation and the possible modification of painful or non-painful symptoms generated by this TMS. The secondary objectives are to assess chronic pain symptoms of these patients quantitatively and qualitatively, to assess expectations of these patients with regard to the performed examinations and to assess their expectations regarding magnetic stimulation performed for therapeutic purposes.

DETAILED DESCRIPTION:
The investigators have therefore developped a questionnaire that will be submitted to all consecutive patients who meet the inclusion criteria and who have given their consent to participate. This questionnaire will be performed in three phases: 1) a few minutes before the realization of evoked potentials and TMS 2) 10 minutes after evoked potentials and TMS 3) two weeks after evoked potentials and TMS (by telephone).

The data collected will be:

- Phase 1 (a few minutes before the explorations): Quantitative assessment of pain Brief Pain inventory Characteristics of pain Analgesic treatments already received and respective efficacy Expectation for diagnostic tests (confirmation/exclusion of diagnosis, …) Expectation for TMS performed for therapeutic purposes (partial/complete recovery, motor/pain symptoms, …)

- Phase 2 (10 minutes after diagnostic explorations and therapeutic TMS): Quantification of pain generated by TMS Quantification of discomfort generated by TMS Change in pain symptoms after TMS Change in motor, sensory or cognitive symptoms after TMS Other side effects of TMS

- Phase 3 (two weeks after TMS, by telephone): Quantitative assessment of pain Brief Pain inventory Quantification of pain generated by TMS Quantification of discomfort generated by TMS Change in pain symptoms after TMS Change in motor, sensory or cognitive symptoms after TMS Other side effects of TMS

ELIGIBILITY:
Inclusion Criteria:

* Patient referred to Avicenne hospital to explore a suspected functional neurological disorder
* Patient able to complete the questionnaire

Exclusion Criteria:

- Lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient referred to Avicenne hospital to explore a suspected functional neurological disorder
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Pain intensity experienced during TMS on a 11-point numerical rating scale (NRS) ranging from 0 (no pain) to 10 (worst possible pain) | 1 hour
  Pain intensity experienced during TMS on a 11-point numerical rating scale (NRS) ranging from 0 (no pain) to 10 (worst possible pain)

SECONDARY OUTCOMES:
Qualitative and quantitative Pain Assessment | 1 hour and 14 days
  Qualitative and quantitative Pain Assessment Brief Pain inventory Pain characteristics
Symptoms post-TMS | 1 hour and 14 days
  Change in pain after TMS. Change in Motor, sensory or cognitive symptoms after TMS. Occured side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- HUPSSD, Bobigny, France

IPD SHARING:
Plan to Share IPD: No